CLINICAL TRIAL: NCT03015519
Title: A Randomized, Double-blind, Placebo Controlled, Multi-center Study to Evaluate the Pharmacokinetics, Safety and Efficacy of Albiglutide for the Treatment of Type 2 Diabetes Mellitus in Pediatric Patients
Brief Title: A Study to Evaluate Pharmacokinetics, Safety and Efficacy of Albiglutide in Pediatric Subjects With Type 2 Diabetes Mellitus
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study did not start recruiting as albiglutide would have been withdrawn from the market prior to study end.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200938
Record Dates: First submitted 2016-12-14; First posted 2017-01-10 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GSK716155; Type 2 diabetes mellitus; albiglutide; safety; pediatric; efficacy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rGLP-1 protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Albiglutide cohort 1: Part A (Experimental): Approximately 12 eligible subjects, aged between 14 to 18 years, will receive a single dose of 30 mg albiglutide post-randomization.
  Interventions: Drug: Albiglutide
- Placebo cohort 1: Part A (Placebo Comparator): Approximately 3 eligible subjects, aged between 14 to 18 years, will receive a single dose of matching placebo post-randomization.
  Interventions: Drug: Placebo
- Albiglutide cohort 2: Part A (Experimental): Approximately 12 eligible subjects, aged between 10 to 14 years, will receive a single dose of 30 mg albiglutide post-randomization.
  Interventions: Drug: Albiglutide
- Placebo cohort 2: Part A (Placebo Comparator): Approximately 3 eligible subjects, aged between 10 to 14 years, will receive a single dose of matching placebo post-randomization.
  Interventions: Drug: Placebo
- Albiglutide: Part B (Experimental): Approximately 120 eligible subjects, aged between 10 to 18 years, will receive albiglutide 30 mg once weekly post-randomization.
  Interventions: Drug: Albiglutide
- Placebo: Part B (Placebo Comparator): Approximately 60 eligible subjects, aged between 10 to 18 years, will receive matching placebo once weekly post-randomization.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Albiglutide — 30 mg of lyophilized albiglutide will be delivered from a prefilled dual chamber glass cartridge (DCC). The pen injector system will deliver 0.5 mL albiglutide as a single subcutaneous injection once a week.
  Arms: Albiglutide cohort 1: Part A; Albiglutide cohort 2: Part A; Albiglutide: Part B
Drug: Placebo — Matching placebo will be delivered from a prefilled dual chamber glass cartridge DCC. The pen injector system will deliver 0.5 mL matching placebo as a single subcutaneous injection once a week.
  Arms: Placebo cohort 1: Part A; Placebo cohort 2: Part A; Placebo: Part B

SUMMARY:
The incidence of Type 2 Diabetes Mellitus (T2DM) is increasing day by day but the treatment options are limited in children and adolescents. Albiglutide, approved for the treatment of T2DM in adult population, is a novel analogue of glucagon-like peptide-1 (GLP-1) with a sufficiently long half-life to permit once a week injection. The study will be conducted in 2 parts: Part A is a single dose pharmacokinetic (PK) study to confirm the dose and safety of albiglutide in pediatric subjects aged 10 to less than 18 years and Part B is a randomized double-blind placebo controlled study to evaluate the safety and efficacy (glycemic control) of albiglutide in the pediatric population. Treatment duration in Part B is 52 weeks (24 weeks double-blind placebo-controlled and 28 weeks open-label during which all subjects will receive albiglutide). Approximately 210 eligible male and female subjects will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Between 10 to less than 18 years of age inclusive at the time of screening.
* Diagnosis of T2DM with HbA1c more than or equal to 7.0% [53 millimole per mole (mmol/mol)] and less than 10.0% (85.8 mmol/mol) assessed at screening. Currently treated with regimen of diet and exercise with or without metformin. Subjects on metformin monotherapy should have been treated for a minimum of 8 weeks prior to randomization on a dose above 1000 milligram per day (mg/day) or prior documented maximum tolerated dose (MTD) less than or equal to 1000 mg/day.
* FPG less than 240 mg/deciliter (dL) at screening.
* Fasting C-peptide more than or equal to 0.8 nanogram per milliliter (ng/mL) at screening.
* Negative central laboratory assays for Glutamic Acid Decarboxylase 65 (GAD-65) and Islet Cell Autoantigen 512 (ICA512) autoantibodies at screening.
* Body weight more than or equal to 30 kilogram (kg) at screening.
* Male subjects will be included. Female subjects who have achieved menarche and are of childbearing potential must be practicing adequate contraception for the duration of participation in the study.
* Signed informed consent of parent or legal guardian and assent as appropriate will be obtained from the child.

Exclusion Criteria:

* Subjects with Type 1 diabetes mellitus or secondary diabetes mellitus (i.e. any type other than T2DM)
* Female subject is pregnant (confirmed by laboratory testing), planning a pregnancy or lactating.
* History of cancer that has not been in full remission for at least 3 years before screening.
* History of thyroid cancer.
* Personal history or family history of thyroid medullary carcinoma or multiple endocrine neoplasia type 2 (MEN2).
* History of pancreatitis or considered clinically at significant risk of developing pancreatitis during the course of the study (e.g. due to symptomatic gallstones).
* Severe gastroparesis within 6 months prior to screening.
* History of significant gastrointestinal (GI) surgery that in the opinion of the investigator is likely to significantly affect upper GI or pancreatic function.
* Have a history of at least one episode of diabetic ketoacidosis (DKA) after receiving anti-diabetic medication.
* Fasting triglyceride level more than 750 mg/dL at screening.
* Serum calcitonin more than 50 picogram (pg/mL) at screening.
* Hemoglobinopathy that may affect determination of HbA1c.
* Uncontrolled hypertension at screening.
* Estimated Glomerular Filtration Rate (eGFR) less than 90 mL/minute/1.73 meter^2 (calculated using the Schwartz equation) at screening.
* ALT more than 2.5x upper limit of normal (ULN) or Bilirubin more than 1.5xULN (isolated bilirubin more than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin more than 35%) at screening.
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
* Current or previous insulin therapy used for more than 4 weeks (continuously) in the 3 months prior to screening.
* Use of a GLP-1receptor agonist at study entry and during the study.
* Any oral diabetic medications, except metformin, at study entry and during the study.
* Use of oral or systemically injected glucocorticoids is generally not allowed within the 3 months before randomization; however, short courses of oral steroids (single dose or multiple doses for up to 7 days) may be permitted provided these cases are discussed with the medical monitor.
* Weight loss medications.
* Antiretroviral drugs.
* Known allergy or serious hypersensitivity reaction to albiglutide or any product components (including yeast and human albumin), any other GLP 1 analogue, insulin, or other study medication's excipients or other contraindications.
* Any other reason the investigator deems the subject to be unsuitable for the study or may interfere with trial compliance (e.g. significant medical or psychiatric history).
* The subject has participated in a clinical trial and has received an investigational product or device within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-08-14 (Estimated); Primary Completion 2020-04-20 (Estimated); Study Completion 2020-04-20 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) of albiglutide: Part A | Up to 28 days post-dose
  Blood samples will be collected prior to dosing at Baseline and following single-dose administration of albiglutide at indicated time points
Maximum Plasma Concentration (Cmax) of albiglutide: Part A | Up to 28 days post-dose
  Blood samples will be collected prior to dosing at Baseline and following single-dose administration of albiglutide at indicated time points.
Apparent clearance (CL/F) of albiglutide: Part A | Up to 28 days post-dose
  Blood samples will be collected prior to dosing at Baseline and following single-dose administration of albiglutide at indicated time points.
Apparent volume of distribution (V/F) of albiglutide: Part A | Up to 28 days post-dose
  Blood samples will be collected prior to dosing at Baseline and following single-dose administration of albiglutide at indicated time points.
Number of subjects with adverse events (AEs): Part A | Up to Week 8 post dose
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. AESI including gastrointestinal events, hypoglycemia, injection site reactions, pancreatitis, medullary thyroid cancer, atrial fibrillation/flutter, and pneumonia etc will also be evaluated.
Change from Baseline in Glycosylated Hemoglobin A1c (HbA1c) at Week 24: Part B | Up to Week 24
  Change in HbA1c values from Baseline will be evaluated at Week 24. The superiority of albiglutide over placebo will be assessed.
Time to reach maximum plasma concentration (tmax) of albiglutide: Part A | Up to 28 days post-dose
  Blood samples will be collected prior to dosing at Baseline and following single-dose administration of albiglutide at indicated time points.
Time to reach half of the maximum plasma concentration (t1/2) of albiglutide: Part A | Up to 28 days post-dose
  Blood samples will be collected prior to dosing at Baseline and following single-dose administration of albiglutide at indicated time points.

SECONDARY OUTCOMES:
Change from Baseline in fasting Plasma Glucose (FPG): Part B | Up to Week 24
  FPG will be assessed as a measure of glycemic control.
Percentage of subjects reaching HbA1c less than 7%: Part B | Up to Week 24
  Subjects reaching HbA1c less than 7% at the end of double-blind phase will be analyzed using logistic regression.
Time to hyperglycemia rescue: Part B | Up to Week 24
  Time to hyperglycemia rescue will be measured at specific timeframe. Addition of or adjustment to metformin will be the first option for rescue therapy.
Number of subjects with AEs, serious adverse events (SAEs): Part B | Up to Week 60
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgement will be categorized as SAE. AESI including gastrointestinal events, hypoglycemia, injection site reactions, pancreatitis, medullary thyroid cancer, atrial fibrillation/flutter, and pneumonia etc will be evaluated.
Number of hypoglycemic episodes: Part B | Up to Week 60
  Hypoglycaemic events as per American Diabetes Association (ADA) criteria: severe hypoglycaemia, documented symptomatic hypoglycaemia, asymptomatic hypoglycaemia, probable symptomatic hypoglycaemia and pseudo hypoglycaemia.
Evaluation of immunogenicity: Part B | Up to Week 60
  Blood samples will be collected at intervals for the determination of anti-albiglutide antibodies.
Change from Baseline in serum calcitonin levels: Part B | Up to Week 52
  Blood samples will be collected to measure serum calcitonin.
Number of subjects with abnormal clinical laboratory parameters: Part B | Up to Week 60
  Hematological, clinical chemistry and urine parameters will be evaluated.
Assessment of Systolic Blood pressure (SBP) and Diastolic Blood Pressure (DBP): Part B | Up to Week 60
  SBP and DBP will be measured in a seated position after at least a 5-minute rest.
Assessment of pulse rate: Part B | Up to Week 60
  Pulse rate will be measured in a seated position after at least a 5-minute rest.
Number of subjects with abnormal growth and development: Part B | Up to Week 52
  Height, weight, tanner stage, menstrual history, sex hormones will be evaluated.
CL/F of albiglutide: Part B | Up to Week 24
  Blood samples will be collected after repeat dose administration of study treatment at indicated time points
V/F of albiglutide: Part B | Up to Week 24
  Blood samples will be collected after repeat dose administration of study treatment at indicated time points
First-order absorption rate constant(Ka): Part B | Up to Week 24
  Blood samples will be collected after repeat dose administration of study treatment at indicated time points
Number of subjects showing covariate relationship between PK and clinical measure of interest: Part B | Up to Week 24.
  The relationship between albiglutide PK parameters and covariates will be evaluated graphically and in the population PK model.
Change from Baseline in Pediatric Quality of Life Inventory (PedsQL) diabetes module total score: Part B | Up to Week 52
  The diabetes module of the PedsQL is a disease specific instrument used to assess the degree of difficulty youth experience with different aspects of everyday living, including treatment adherence and barriers, diabetes-related worries, and communication with others about diabetes. Scores range from 0 to 100, with a higher PedsQL scores indicating better levels of functioning and quality of life (QOL).
Change from Baseline in Children's Depression Inventory 2 Self Report Short Version [CDI 2: SR(S)] | Up to Week 52
  The CDI 2: SR(S) is a revision of the Children's Depression Inventory and is used to evaluate depressive symptoms in children and adolescents. The CDI 2: SR(S) Form contains 12 items and the domains include emotional problems and functional problems, with additional subscales of negative mood/physical symptoms, negative self-esteem, interpersonal problems and ineffectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Morehead City, North Carolina
  - GSK Investigational Site, El Paso, Texas